CLINICAL TRIAL: NCT05169255
Title: Long Term Antibiotics Study
Brief Title: Impact of Prolonged Antibiotic Therapy on Commensal Microbial Community Gene Expression.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, David Pride, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 121456
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Two parallel groups with placebo versus antibiotics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin (Experimental): 24 participants received azithromycin for 3 or 7 days
  Interventions: Drug: Antibiotic administration
- Amoxicillin (Experimental): 24 participants received amoxicillin for 3 or 7 days
  Interventions: Drug: Antibiotic administration

INTERVENTIONS:
Drug: Antibiotic administration — Individuals received either azithromycin or amoxicillin for 3 or 7 days

SUMMARY:
Antibiotics are a mainstay of life-saving interventions used frequently in medical practice to combat infections. These medications not only target the pathogenic bacteria for which they are prescribed but also function against commensal bacterial communities that inhabit the gut, skin, and oropharynx. The role that these native bacterial communities play in normal host function, such as in nutrition and host immunity, is only beginning to be explored, as are the changes in the communities and their function as a result of various alterations of antibiotic use. Short courses of antibiotics have been shown to affect the diversity of native bacterial communities, and to affect the abundance of antibiotic resistance genes present. For example, use of clindamycin in human subjects for 7 days has been demonstrated to result in persistent clindamycin resistance for months or years. The impact of prolonged antibiotic therapy on the host microbiome including both those organisms present and the diversity of antibiotic genes has not been studied, and we have very little understanding of the longitudinal effects of antimicrobial therapy on the genetic repertoire present in human microbial communities. In this study, we will examine changes in the microbiota as well as frequency of antibacterial resistance genes harbored in skin, saliva, and colonic microbiomes longitudinally in subjects on prolonged antimicrobial therapy, as well as household members of the person on antibiotic therapy. Previously well patients with minimal prior antibiotic exposure will be enrolled upon diagnosis of an infection requiring long-term antibiotic therapy, such as osteomyelitis or prosthetic joint infection, prior to starting antibiotic therapy. We will examine the microbiota of the skin, saliva, and gut prior to antibiotics as well as the frequency of antibiotic resistance genes harbored within these microbial communities. We will compare microbial communities and antibiotic resistance gene frequencies before, during and after prolonged course of antibiotics in patients on antibiotics. We will also look for alterations that occur among microbiomes or antibiotic resistance genes among household members of people on antibiotics.

DETAILED DESCRIPTION:
Commensal flora are thought to play important roles in maintaining human health. Bacterial communities and the antibiotic resistance genes harbored within them are likely altered by selective pressure imposed by antibiotic use in clinical settings. Perturbations to the endogenous microbial communities as a result of antibiotic use may have a significant impact on the microbiome and the antibiotic resistance genes carried within. We aim to study how microbial communities are altered by prolonged antibiotic therapy using metagenomics techniques. In addition to measuring the diversity of bacterial genotypes present, we plan to characterize the repertoire of antibiotic resistance genes in human subjects exposed to prolonged courses of antibiotics. We also will measure the effect of environment on the antibiotic resistance repertoire of human microbial communities by assessing antibiotic genes present in subjects that reside in the same household compared to other subjects.

Aim 1: To improve our understanding of the effects of prolonged antibiotic courses on native bacterial communities of human skin, mouth, and colon during and after therapeutic courses of antibiotics. We will look at alterations in bacterial diversity within these communities in quantity as well as quality (how classes of bacteria are altered) using metagenomics.

Aim 2: To improve our understanding of effects of prolonged antibiotic use on the presence of antibiotic resistance genes in the human microbiome over time. We will follow presence and diversity and quantity of antibiotic resistance genes present in commensal bacterial communities longitudinally before, during, and following prolonged antibiotic courses.

Aim 3: To assess whether the bacterial communities present in members of the same household are changed as a result of environmental influences rather than direct antibiotic administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75
* Capacity to give consent, provide samples, and follow-up at routine clinic appointments

Exclusion Criteria:

* Antibiotic use (outside of 72 hour period prior to diagnosis or peri-operative short course) within the 3 months prior to enrollment
* Unable to provide consent or samples
* immunocompromised conditions such as HIV/AIDS, SLE, organ or bone marrow transplant recipient, on immunosuppressants for autoimmune disease, genetic disorders such as cystic fibrosis that may result in substantial alteration in colonized community.
* inability to provide 3mL of saliva without stimulation
* critical illness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12-07 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2016-04-22 (Actual)

PRIMARY OUTCOMES:
Microbiome | 6 months
  Individuals received 3 or 7 days of antibiotics and were followed for 6 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ly M, Jones MB, Abeles SR, Santiago-Rodriguez TM, Gao J, Chan IC, Ghose C, Pride DT. Transmission of viruses via our microbiomes. Microbiome. 2016 Dec 2;4(1):64. doi: 10.1186/s40168-016-0212-z. PMID 27912785
- [Result] Abeles SR, Jones MB, Santiago-Rodriguez TM, Ly M, Klitgord N, Yooseph S, Nelson KE, Pride DT. Microbial diversity in individuals and their household contacts following typical antibiotic courses. Microbiome. 2016 Jul 30;4(1):39. doi: 10.1186/s40168-016-0187-9. PMID 27473422
- [Derived] Chopyk J, Cobian Guemes AG, Ramirez-Sanchez C, Attai H, Ly M, Jones MB, Liu R, Liu C, Yang K, Tu XM, Abeles SR, Nelson K, Pride DT. Common antibiotics, azithromycin and amoxicillin, affect gut metagenomics within a household. BMC Microbiol. 2023 Aug 2;23(1):206. doi: 10.1186/s12866-023-02949-z. PMID 37528343